CLINICAL TRIAL: NCT07201090
Title: Effects and Implementation of a Brief Version of Parent-Child Interaction Therapy, Supplemented by Videos and Virtual Reality-films
Brief Title: Effects and Implementation of a Brief Version of Parent-Child Interaction Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Pia Enebrink, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-08744-01
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Conduct Disorders in Children; Disruptive Behavior; Oppositional Defiant Disorder
Keywords: Parent training; Parent-Child Interaction Therapy; Virtual reality
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Parent-Child Interaction Therapy with videos and virtual reality (360-degree VR)-films (Experimental): 10 sessions of Parent-Child Interaction Therapy (PCIT), supplemented with brief role-modeling videos of parenting skills, provided through an online project platform, and virtual reality (360-degree VR)-films shown during treatment sessions.
  Interventions: Behavioral: Brief Parent-Child Interaction Therapy with videos and virtual reality (360-degree VR)-films

INTERVENTIONS:
Behavioral: Brief Parent-Child Interaction Therapy with videos and virtual reality (360-degree VR)-films — 10 sessions of PCIT delivered by trained psychologists, supplemented with videos and 360-degree VR-films
  Sessions follow the standard PCIT structure, with an initial phase focused on child-directed interaction, followed by a second, modified phase, focused on parent-directed interaction.
  To support skill learning, families are provided with digital materials including conventional video modules at home and 360-degree virtual reality (VR) films. The VR films are shown during two sessions at the clinic. Additional videos are available online through a platform for parents to view and practice between sessions. These tools allow parents to rehearse skills flexibly in their home environment and reinforce the in-session training.
  Other Names: Brief PCIT-VR

SUMMARY:
The aim of this study is to evaluate the effects and feasibility of a shortened version of Parent-Child Interaction Therapy (PCIT), supplemented with video vignettes of parenting skills and 360-virtual reality (VR)-films for parents of children aged 2-7 years with disruptive behavior problems. The main questions the study aims to answer, using a Single-Case Experimental Design, are:

1. How feasible and acceptable is the implementation of brief PCIT-VR in Sweden?
2. What are the preliminary effects of brief PCIT-VR?
3. How do parents and clinicians experience brief PCIT-VR?

Families at child and adolescent psychiatry clinics will receive up to 10 PCIT sessions. Caregivers complete quantitative assessments before, during, after treatment, and at 6-months follow-up, and are asked to participate in interviews after PCIT. Feasibility and acceptability of brief PCIT VR is evaluated, as well as effectiveness outcomes, including changes in child disruptive behavior and parenting skills. Within-group analyses will examine trends in outcome measures over time.

DETAILED DESCRIPTION:
BACKGROUND:

Persistent and clinically significant behavior problems are associated with long-term negative outcomes if left untreated. Early and effective interventions are critical for children's development and to reduce long-term societal costs.

Parent training programs are the most effective evidence-based interventions for children under 12 years with externalizing behavior problems. Parent-Child Interaction Therapy (PCIT) is one of the most rigorously evaluated programs for children aged 2-7 years. PCIT is distinctive in that it uses live coaching, where the therapist guides parents in real time as they interact with their child. Several meta-analyses demonstrate large effects of PCIT in reducing child disruptive behavior and improving parenting skills.

However, both the length of PCIT treatment and dropout rates remain challenges. The PCIT protocol often requires 15-25 sessions, and high attrition rates have been reported in routine care. Promisingly, research suggests that PCIT can still be effective when families end treatment early or when time-limited PCIT protocols are used. Further evaluations are needed to understand how effectiveness in briefer treatment formats can be maintained.

Using films and videos for parenting skills modelling, and virtual reality (VR) for practice may enhance skill learning and allow parents to continue practicing outside therapy sessions. VR can provide realistic training opportunities, enabling parents to observe and rehearse parenting skills. A study in the Netherlands has used VR in PCIT with promising results.

This study will implement and evaluate a time-limited (shortened) PCIT format combined with VR and film-based components (brief PCIT-VR). By limiting treatment to 10 sessions and supplementing with these pedagogical tools, the intervention aims to balance effectiveness with feasibility.

PURPOSE AND RESEARCH QUESTIONS:

This study will evaluate preliminary effects, aspects of feasibility, and experiences with brief PCIT-VR.

Research questions:

1. How feasible and acceptable is the implementation of brief PCIT-VR in Sweden?
2. What are the preliminary effects of brief PCIT-VR?
3. How do parents and clinicians experience brief PCIT-VR?

METHOD:

This study will use a Single-Case Experimental Design (SCED).

Participants will be families including parents of children aged 2-7 years who present with disruptive behavior problems according to >114 on the Eyberg Child Behavior Inventory (ECBI). Families will be recruited through child and adolescent psychiatry clinics in Sweden. Clinicians working at these clinics will provide initial information about the study orally and in writing. Parents who express interest will be directed to an online portal where they receive written information. Both legal guardians provide written informed consent before participation. Parents fill out the ECBI to inform whether they meet inclusion criteria. A person from the research group contacts the family to provide more information and inform about inclusion or exclusion. If families are included, they are provided with login to a platform where they respond to weekly measurements, baseline/post treatment measurements, and during the treatment phase have access to video vignettes illustrating parenting skills. Parents will also have access to brief virtual reality-films at the clinic together with the therapist during two PCIT-sessions.

The study consists of three main phases: baseline, treatment, and follow-up. During the baseline phase (before treatment starts during approximately three weeks) and during the treatment phase, parents complete weekly questionnaires. In the middle of the treatment, parents respond to a longer measurement (ECBI). Before and after treatment, a larger battery of questions are administered (pre-, post- treatment, and 6-month follow-up assessments).

Each week during PCIT, parents are given access to a new module in the online platform with video vignettes of parenting skills, supplementing the session. The treatment phase involves up to 10 PCIT sessions. Semi-structured qualitative interviews will be conducted with both parents and clinicians after treatment to explore experiences, feasibility, and acceptability.

SAMPLE SIZE CALCULATION:

We aim to include a target of 15 families (approximately 15-30 parents), in line with SCED-study standards and similar SCED studies conducted internationally.

ANALYSES:

Quantitative data will be analyzed using visual inspection of weekly SCED graphs and statistical methods such as percent change calculations, Reliable Change Index analyses, and repeated-measures analyses of variance (ANOVA). Benchmarking will be used to compare outcomes with those from longer PCIT trials reported in the literature. Qualitative interview data will be analyzed thematically to identify key themes regarding feasibility, acceptability, and barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 2-7 years
* Elevated disruptive behavior (ECBI score >114)
* Parent speaks Swedish or English

Exclusion Criteria:

* Child or family requiring more urgent intervention
* Parent condition that prevents VR use (e.g., epilepsy, severe migraine, adverse VR experiences)

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from screening in parent-ratings of child behavior problems on the Eyberg Child Behavior Inventory (ECBI) - Intensity scale | Screening (at inclusion), pre-treatment (treatment phase week 0), mid treatment (treatment phase week 6), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  Measures frequency of externalizing behaviors in children. The scale includes 36 items which are rated on a 7-point-scale (1 to 7). The total scale sum ranges from minimum 36 to a maximum sum of 252. Higher score indicates more disruptive behavior problems.
Mean change from screening in parent-ratings of child behavior problems on the Eyberg Child Behavior Inventory - Problem scale | Screening (at inclusion), pre-treatment (treatment phase week 0), mid treatment (treatment phase week 6), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  Measures externalizing behaviors in children. The scale includes 36 items which are rated yes/no (1-0), indicating whether the behavior is experienced as problematic. Minimum summary score is 0, maximum score is 36. Higher score indicates more disruptive behavior problems.
Change from baseline phase to treatment phase in weekly reported disruptive behavior | Weekly throughout baseline phase (baseline phase week 1-4) and treatment phase (treatment phase week 1-10).
  Three weekly questions on disruptive behavior rated on an 8 point scale from 0-7. Minimum summary score is 0, maximum score is 21. Higher score indicates more disruptive behaviors.

SECONDARY OUTCOMES:
Mean change from pre-treatment in parent-rated callous unemotional behaviors on the Inventory of Callous Unemotional traits (ICU) scale | Pre-treatment (treatment phase week 0), post-treatment (treatment phase week 10)
  The 12 item version of the Inventory of Callous Unemotional scale measures perceived callous or unemotional behaviors. The scale consists of 12 items rated on a 4-point Likert scale from 0 to 3. Total scores range from 0 to 36, with higher scores indicating higher levels.
Mean change from pre-treatment in parent-rated stress on the Perceived Stress Scale (PSS) | Pre-treatment (treatment phase week 0), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  The 10 item Perceived Stress Scale measures perceived stress on a 5-point Likert scale scored 0-4 (minimum scale value is 0, maximum is 40). Higher scores indicate more stress.
Mean change from pre-treatment in parent-rated parenting behaviors on the Parenting Young Children (PARYC) - frequency scale | Pre-treatment (treatment phase week 0), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  A 21 item rating scale completed by parents, measuring parenting behaviors and strategies. Parents rate the frequency of parenting strategies/activities on a scale scored 1-5 (ranging between 21-105). Higher values represent using positive parenting strategies more frequently.
Mean change from pre-treatment in parent-rated parenting behaviors on the Parenting Young Children (PARYC) - problem scale | Pre-treatment (treatment phase week 0), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  A 21 item rating scale completed by parents, measuring parenting behaviors and strategies. Parents indicate whether they find performing the parenting strategy/activity problematic (yes/no; rated 1-0), with a summary score ranging between 0-21. Higher values reflect greater parenting challenges.
Change from baseline phase to treatment phase in weekly reported warmth and relationship quality | Weekly throughout baseline phase (baseline phase week 1-4) and treatment phase (treatment phase week 1-10).
  Four weekly questions on warmth and relationship-enhancing behaviors (playing, doing nice things, positive attention and affection). Rated on a 7 point scale from 0-6. Minimum summary score is 0, maximum summary score is 24. Higher scores indicate higher levels of warmth and relationship-enhancing behaviors.
Change from baseline phase to treatment phase in weekly reported parental anger | Weekly throughout baseline phase (baseline phase week 1-4) and treatment phase (treatment phase week 1-10).
  One weekly question of whether parents have felt upset with or angry at their children. Rated on a 7 point scale from 0-6. Higher score indicates more frequent experiences of anger.
Change from baseline phase to treatment phase in weekly reported emotion regulation | Weekly throughout baseline phase (baseline phase week 1-4) and treatment phase (treatment phase week 1-10).
  If parents report being angry at least once across the past week, two follow-up questions inquire about how parents handled the situation. These items are rated on a 6 point scale scored 0-5. Summary score ranges between 0 and 10. Higher scores indicate more frequent instances of remaining calm.
Change from baseline phase to treatment phase in weekly reported consistent parenting | Weekly throughout baseline phase (baseline phase week 1-4) and treatment phase (treatment phase week 1-10).
  One item assesses whether parents have been consistent with holding on to rules despite repeated requests from their children. Responses are rated on a 6 point scale (0-5), with higher scores indicating greater consistency.
Mean change from baseline in parental emotion regulation on the Parent Emotion Regulation Scale | Pre-treatment (treatment phase week 0), post-treatment (treatment phase week 10), and at 6-months follow-up (6 months from pre-treatment assessment)
  Parental emotion regulation will be measured with the Parent Emotion Regulation Scale. The 20 items are scored on a 5-point scale (1 to 5). A total summary score ranges between 20 and 100, where a higher score indicates better regulation of emotions.

OTHER OUTCOMES:
Post treatment satisfaction on the Therapy Attitude Inventory | Post-treatment (treatment phase 10 weeks)
  Parent-rated therapy satisfaction is evaluated with the Therapy Attitude Inventory, which includes 10 items, each rated between 1 to 5. Total sum ranges between 10-50, where a higher score indicates more satisfaction with treatment.
Parental experiences of the treatment explored through individual qualitative interviews | Post-treatment (treatment phase 10 weeks)
  Qualitative interviews will explore parent's experiences of participating in the treatment and of using parental strategies, and includes questions about experienced effectiveness, feasibility, satisfaction. Three questions target helpfulness, relevance and usefulness, and are rated 0-10. Total sum ranges between 0-30, with higher scores indicating greater levels of usefulness.
Clinician experiences of the treatment explored through individual qualitative interviews | Post-treatment (treatment phase 10 weeks)
  Qualitative interviews will explore clinicians' experiences of the treatment and includes questions about experienced effectiveness, feasibility, satisfaction.
Caregiver: Background information | First weekly assessment (baseline phase week 1)
  A few questions on caregiver and child background.
Parent reported satisfaction with the online video modules | Weekly during treatment phase (up to 10 weeks)
  Caregivers report satisfaction with the videos in each online module through 4 questions rated on a 5 point scale scored 1-5 (total summary score is minimum 4, maximum 20). Higher score indicates greater satisfaction.
Parent-reported experience with the online modules | Weekly during treatment phase (up to 10 weeks)
  Caregivers report in free text their experiences with online modules, e.g., if something was difficult to understand or was missing.
Clinician-rated manual adherence and family alliance | Weekly during treatment phase (up to 10 weeks)
  5 weekly questions to clinicians on manual adherence and experienced alliance with families. Rated on an 11 point scale from 0 to 10 (total weekly summary score is minimum 0, maximum is 50). Higher score indicates greater adherence and alliance.
Parent completion of online modules and treatment sessions | Weekly during treatment phase (up to 10 weeks)
  The number of modules completed are assessed through data from the online platform and completed sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Enebrink, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Solna
  - Region Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: No